CLINICAL TRIAL: NCT02497833
Title: Effect of Retinoic Acid Supplementation on the HDL-Associated Paraoxonase 1 Activity in Subjects With Hypercholesterolemia: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Retinoic Acid Supplementation and Subjects With Hypercholesterolemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Di Li, Doctor of Medicine, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZXYZM-2
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Tretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): the participants in this arm are instruted to consume placebo capsules
  Interventions: Other: placebo
- treatment (Experimental): the participants in this arm are instruted to consume retinoic acid capsules
  Interventions: Dietary Supplement: retinoic acid

INTERVENTIONS:
Dietary Supplement: retinoic acid — During the trial period, the participants are instructed to consume retinoic acid capsules twice daily (30 min after breakfast and supper).The retinoic acid capsules provided a total daily intake of 10 mg of retinoic acid.
  Arms: treatment
Other: placebo — During the trial period, the participants are instructed to consume placebo capsules twice daily (30 min after breakfast and supper).The placebo capsules are composed of starch and pigment.
  Arms: control

SUMMARY:
The aim of the study is to investigate the effects of retinoic acid on the HDL-PON1 activity and cholesterol efflux capacity in hypercholesterolemic subjects.

DETAILED DESCRIPTION:
Paraoxonase 1 (PON1), an enzyme associated with high-density lipoprotein, is reported to have antioxidant and cardioprotective properties. And all-trans-retinoic acid revealed the ameliorating atherosclerosis effects in many reports.There maybe some correlations between retinoic acid and PON1 activity and the study aim to prove it.

ELIGIBILITY:
Inclusion Criteria:

* subject has a fasting total cholesterol concentration between 200 and 310mg/dl.
* subject is between 25 and 65 years of age, inclusive.
* subjects' BMI is between 18.5 kg/m2 and 35 kg/m2.

Exclusion Criteria:

* subject that is pregnant.
* subject that has coronafy artery desease, diabetes mellitus, thyroid disorders, mental disorder, cancer, cirrhosis, renal disease and hepatic desease.
* subject that has had operation less than six months prior to screening visit.
* subject that is smoking.
* subject uses any drugs that could influence the measurement of lipid paramerters or inflammatiory makers.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
PON1 activity | changes from baseline in PON1 activity at 12 weeks
  PON1 activity is assayed in HDL isolated from plasma of subjects from the placebo and retinoic acid groups by using UV spectrophotometry in a 96-well plate format using phenyl acetate or paraoxon as substrates.

SECONDARY OUTCOMES:
Lp-PLA2 activity | changes from baseline in Lp-PLA2 activity at 12 weeks
  Lp-PLA2 activity in apoB-depleted plasma after the sedimentation of all apoB-containing lipoproteins with dextran sulfate-magnesium chloride is determined using the trichloroacetic acid precipitation procedure using 2-thio platelet-activation factor as a substrate.

OTHER OUTCOMES:
cholesterol efflux capacity | changes from baseline in cholesterol efflux capacity at 12 weeks
  The cholesterol efflux capacity of the two groups at baseline and after intervention is quantified by a modified method with J774 mouse macrophages. After plated and radiolabeled with 3H-cholesterolper, J774 macrophages are incubation with cAMP and apoB-depleted serum successively. Liquid scintillation counting is used to quantify the efflux of radioactive cholesterol from the cells.

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Study Director — Sun Yat-sen University
Locations (1):
- Guangdong Provincial Key Laboratory of Food, Nutrition and Health, Department of Nutrition, School of Public Health, Sun Yat-Sen University (Northern Campus), Guangzhou, Guangdong, China